CLINICAL TRIAL: NCT01480375
Title: A 3D Navigation Technology for Improved TRUS Prostate Biopsy
Brief Title: A Novel 3D Navigation Technology for Improved TRUS Prostate Biopsy
Acronym: NaSBxP01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UC Care, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0053-11-BNZ
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
Keywords: prostate cancer detection; prostate biopsy; 3d navigation; trans rectal ultrasound
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Navigo™ and Smartbx™ system. (Experimental): all biopsy cores were handled using the Smartbx™ system. part of the procedures were performed with both Navigo™ and Smartbx™ system.
  Interventions: Device: Smartbx™ system.
- standard method (No Intervention): all biopsy cores were handled using standard method - shaking the biopsy needle into formalin vial. no navigation system.

INTERVENTIONS:
Device: Smartbx™ system. — The SmartBx™ system semi-automated downloads the biopsy cores from the biopsy needle onto a designated cassette which integrates into the routine pathology lab processing. The core is downloaded in an oriented and straightened fashion while preserving core fragments in its original locations relative to the needle notch.
  Arms: Navigo™ and Smartbx™ system.

SUMMARY:
he most common method for performing a prostate biopsy procedure is the ultrasound guided transrectal procedure. The information obtained from the standard prostate biopsy is deficient and even misleading. Cancers can be missed on initial and even in repeated biopsy. Moreover, the detection of a tumor cannot predict accurately the tumor size and location1. It was proven that the exact location of the obtained cores, even in an initial biopsy, can influence the cancer detection rate2.

An imaging tool that will enable a three-dimensional navigation in the prostate volume and selecting biopsy locations in view of previous core taken will allow building a "tumor map" '(i.e. detecting tumor size and location). By mapping the prostate cancer an adequate treatment can be chosen while avoiding over or insufficient treatment.

However, to be able to produce an accurate mapping of the malignant tissue, a complementary optimized pathology method should be also implement in addition to the navigation system, it has been shown that a pre-embedding procedure that keeps the specimen orientation, unfolding, unity, and location along the needle notch improves the histological yield and hence the cancer detection rate3.

The NaviGo™ Workstation (hereafter the NaviGo™ Workstation or the NaviGo™ System) allows physicians to see the prostate gland together with the biopsy sites in a three dimensional (3D) view, modeled from two dimensional (2D) images. The NaviGo™ Workstation was designed as an adjunct to standard of care procedures, to work with standard rectal ultrasound probes, and to be incorporated side by side with the techniques currently employed. No change to the current employed procedures and techniques is required or suggested. In complementary to the Navigo system a system for semi-automatic download of prostate biopsy cores which keeps the orientation, unfolding and unity of the sample was developed to increase the pathology utility.

The study objective is to evaluate the contribution of the Navigo™ system, an aiding navigation tool for TRUS prostate biopsy, to an increase in the prostate cancer detection ability.

DETAILED DESCRIPTION:
Introduction Prostate biopsy is a procedure in which small samples are removed from a man's prostate gland to be later tested for the presence of cancer. It is typically performed when the scores from a PSA blood test rise to a level that is associated with the possible presence of prostate cancer.

The most common method for performing a prostate biopsy procedure is the ultrasound guided transrectal procedure. The information obtained from the standard prostate biopsy is deficient and even misleading. Cancers can be missed on initial and even in repeated biopsy. Moreover, the detection of a tumor cannot predict accurately the tumor size and location1. It was proven that the exact location of the obtained cores, even in an initial biopsy, can influence the cancer detection rate2.

An imaging tool that will enable a three-dimensional navigation in the prostate volume and selecting biopsy locations in view of previous core taken will allow building a "tumor map" '(i.e. detecting tumor size and location). By mapping the prostate cancer an adequate treatment can be chosen while avoiding over or insufficient treatment.

However, to be able to produce an accurate mapping of the malignant tissue, a complementary optimized pathology method should be also implement in addition to the navigation system, it has been shown that a pre-embedding procedure that keeps the specimen orientation, unfolding, unity, and location along the needle notch improves the histological yield and hence the cancer detection rate3.

The NaviGo™ Workstation (hereafter the NaviGo™ Workstation or the NaviGo™ System) allows physicians to see the prostate gland together with the biopsy sites in a three dimensional (3D) view, modeled from two dimensional (2D) images. The NaviGo™ Workstation was designed as an adjunct to standard of care procedures, to work with standard rectal ultrasound probes, and to be incorporated side by side with the techniques currently employed. No change to the current employed procedures and techniques is required or suggested. In complementary to the Navigo system a system for semi-automatic download of prostate biopsy cores which keeps the orientation, unfolding and unity of the sample was developed to increase the pathology utility.

OBJECTIVE AND RATIONALE Study objective Evaluate the contribution of the Navigo™ system, an aiding navigation tool for TRUS prostate biopsy, to increase the prostate cancer detection ability.

Rationale

The Navigo™ system is a noninvasive navigation tool that produces on line 3D model of the prostate that assist the physician to navigate in the prostate volume during the biopsy procedure without changing the imaging system or the biopsy routine whatsoever. The ability to create a 3D model of the prostate and accurately and evenly position the biopsy needle will enable a more accurate biopsy and better analysis of the procedure and the pathological results, hence it might improve the clinical outcomes and may lead to new treatments/diagnostic strategies.

DEVICE DESCRIPTION AND INTENDED USE

The NaviGo workstation is used as an adjunct to the ultrasound imaging and biopsy procedures of the prostate gland. When operated in conjunction with the standard equipment in a TRUS guided prostate biopsy procedure, the NaviGo™ software may be used for the following:

* To assist the physician by transfer and display of ultrasound images on the workstation screen;
* Build display and manipulate a 3D model of the prostate on screen;
* Archiving the ultrasound images and the 3D model;
* Providing data management solutions;
* Tracking, displaying and recording of the biopsy needle trajectory location in real time.

The NaviGo™ Workstation is designed to work with standard transrectal ultrasound system without changing or interfering with the physician's flow of work. The ultrasound images are displayed on the ultrasound system, and the information provided by the NaviGo provides supplementary information to the physician during the procedure. The NaviGo™ Workstation connects to the video output of the ultrasound system and tracks the ultrasound probe's position using an off-the-shelf electromagnetic tracking system consisting of two sensors, one on the ultrasound probe (at the base/ non invasive part of the probe) and the other on the patient's back, a transmitter placed beneath the patient mattress, a processing unit, a laptop computer and the workstation screen. Figure 1 below presents a general view of the NaviGo™ Workstation.

The NaviGo™ system is an aiding tool in the management of prostate biopsy procedure. The NaviGo™ system allows prostate biopsy tracking, recording, and management solution. The NaviGo™ system is designed to assist the physician in performing prostate biopsy procedures by displaying a 3D model with real-time tracking and recording of the biopsy needle location. The device includes means to compensate for patient body and prostate motion at any time during the procedure. The 3D model can be rotated, manipulated and displayed in the physician's preferable choice.

The Navigo™ system is intended to record and display in 3D the biopsy procedure of any patient undergoing a prostate trans-rectal biopsy. The Navigo™ system is intended to record all the data from the initial scan, the volume measurements, and the biopsy needle insertion. All the images are saved and can be reviewed in post analysis, the needle location can be updated according to the physician's marking on the recorded ultrasound image and the pathology results will be displayed in color on the 3D model.

In post procedure, the physician defines the boundaries of the prostate on selected ultrasound images and a 3D model of the prostate is displayed with all recorded biopsy specimens' locations displayed in the prostatic volume. The physician will be able to examine in post analysis the scattering quality of the biopsy specimens in the prostatic volume and update the pathology results.

Summary of features/capabilities incorporated in the NaviGo™ Workstation.

1. Patient data management (recording, retrieval, off-line analyses and addition of biopsy results).
2. Contour-based 3D model of the prostate (surface rendering).
3. Real-time tracking of the needle trajectory - the trajectory is displayed on the 3D model.
4. Recording of biopsy locations - using operator supplied information regarding where biopsies were obtained, a 20mm long mark is provided on the bottom part of the 3D model (where the trajectory crossed the 3D model), with each mark numbered and linked to the relevant saved US image.
5. Prostate volume calculation and measurement - a 3D model is displayed with volume calculation, and 2D measurement capabilities (point to point inside the model) are available.
6. Off line procedure planning - on the previous acquired 3D model with the updated pathology results the physician can schematically place future biopsy locations.
7. Pathology results management and display - update of the pathology results to the 3D model and a color display according to the severity of the results.
8. Procedure report - automatically generated by the end of each procedure in an HTML format. The report can also be saved to an external memory device or viewed at a later time.

METHODS AND PROCEDURES Study Design

1. The study is an open prospective study.
2. The trans-rectal ultrasound guided prostate biopsy procedure will be conducted according to the standard 12 biopsy scheme.
3. In addition to normal procedure set up, there will be Electromagnetic flat transmitter under the patient's mattress, 2 externally attached sensors and the Navigo™ system stand including a laptop computer and the workstation screen (detailed in appendix A - User's Manual).
4. Following the initial prostate scanning and the standard volume measurements done by the physician, a 3D on-line model will be produced as supplementary information to the B-mode standard image. The physician will navigate and determine the biopsy position using the standard B-mode ultrasound image and the 3D prostate on- line model, both shown on the working station screen.
5. The biopsy samples obtained will be placed straightened in a designated pathology cassette or a kit for the orienting of biopsies, constituted from nitrate cellulose filtering membranes. (See appendix B, C).
6. Patient details, core locations in the prostate volume are saved for future analysis and planning.
7. The data obtained in these experiments will be compared to a retrospective data from a comparable cohort of patients who went through standard procedures with the same biopsy scheme. (The control cohort will be chosen to have similar patient's characteristics- age, PSA level).

End points

* Cancer detection rate (via pathology) compared with a control group- standard 12 biopsy from retrospective data.
* Analysis of positive cores distribution in the prostate volume.
* Detection rate vs. PSA level.

SUBJECT RECRUITMENT

Study population will be recruited from the pool of patients who are scheduled for standard trans-rectal biopsy procedure

POTENTIAL BENEFITS TO THE PATIENTS

The Navigo™ system is a navigation aiding tool which assists the physician to navigate in the prostate volume. The physician can locate the biopsy core according to the desired biopsy scheme. The physician can see on-line the location of the previous cores obtained, and thus gaining the advisable dispersing of the cores and avoiding an overlap between adjacent cores. Core positions are saved for post procedure analysis and future planning. Therefore the patient can gain from an accurate positioning of the biopsy cores, which may increase the cancer detection rate in the current biopsy and produce baseline information for future procedures.

POTENTIAL RISKS TO THE PATIENTS

The Navigo™ system is an aiding tool that does not require any change in the procedure performed today and doesn't come instead of the B-mode ultrasound, but works in parallel to it, to add 3D information. The various components do not come in direct contact with the patient or the physician and the computer and 3D tracking system are well within the required safety protocols. Hence, there is no risk to the patients.

The 3D tracking system is approved by the FDA for medical use and is classified as Type CF which is the most stringent classification, being required for those applications where the applied part is in direct conductive contact with the heart or other applications as considered necessary. The 3D tracking system is also part of an approved Helsinki trial in Bnei-Zion hospital (monitoring of the birth progress, trial initiated by Dr. Yoav Paltieli) Adverse effects, any pain or discomfort to the patients are not expected according to the accumulated experience gained in a series of preliminary experiments preformed on 30 patients with the Navigo™ system in Bnei-Zion as part of a Helsinki trail (0101-10-BNZ). The system is also approved to be used in Haemek medical center (Helsinki number, 0018-11) and Meir medical center (?). Therefore, in view of the above mentioned information there is no risk to the patients and to the users.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Planned for trans-rectal prostate biopsy
* Signed informed consent

Exclusion Criteria:

* Patient's unwilling to participate
* Patients with metal prosthetics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2011-09-22 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
increased prostate cancer detection rate | 30 days
  prostate cancer detection rate would be compared to that of a retrospetive cohort of patients who underwent prostate biopsy without the Navigo device.

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Nativ, Prof., Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion medical center, Haifa, Israel